CLINICAL TRIAL: NCT02747979
Title: The Effect and Safety of Combination Hemodialysis and Hemoperfusion on Severe Renal Osteopathy and Itching in Uremia Patients
Brief Title: The Effect and Safety of Hemodialysis and Hemoperfusion on Severe Renal Osteopathy and Itching in Uremia Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-HD+HP
Record Dates: First submitted 2015-05-21; First posted 2016-04-22 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Hyperparathyroidism; Refractory Pruritus; Ostalgia; Insomnia
Keywords: hemodialysis; hyperparathyroidism; refractory pruritus; ostalgia; insomnia; CVD incidence; life quality
MeSH Terms: conditions — Hyperparathyroidism; Pruritus; Sleep Initiation and Maintenance Disorders | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- hemodialysis+hemoperfusion (HA330) (Experimental): Combination of hemodialysis and hemoperfusion (HA330) therapy All subjects in the study phase will receive hemodialysis plus hemoperfusion(HA330) treatment once per week, and regular hemodialysis treatment in the remaining two sessions.
  Interventions: Other: hemodialysis only; Other: hemodialysis plus hemoperfusion(HA330)
- hemodialysis+hemoperfusion (HA130) (Experimental): Combination of hemodialysis and hemoperfusion (HA130) treatment All subjects in the study phase will receive hemodialysis and hemoperfusion(HA130) treatment once per week, and regular hemodialysis treatment in the remaining two sessions.
  Interventions: Other: hemodialysis only; Other: hemodialysis plus hemoperfusion(HA130)
- hemodialysis only (Active Comparator): hemodialysis only All subjects in the study phase will receive regular hemodialysis treatment three times per week.
  Interventions: Other: hemodialysis only

INTERVENTIONS:
Other: hemodialysis only — hemodialysis treatment only
Other: hemodialysis plus hemoperfusion(HA330) — combination of hemodialysis and hemoperfusion (HA330) treatment
  Arms: hemodialysis+hemoperfusion (HA330)
Other: hemodialysis plus hemoperfusion(HA130) — combination of hemodialysis and hemoperfusion (HA130) treatment
  Arms: hemodialysis+hemoperfusion (HA130)

SUMMARY:
A prospective, randomized, controlled open clinic trial to evaluate the effect and safety of combination of conventional hemodialysis(HD) and hemoperfusion(HP) on middle molecules removal and complications improvement in long-term maintenance hemodialysis (MHD) patients.

There are two phases of study for each subject. Phase 1 (screening phase). During this phase, each potential subject will be evaluated to determine if he/she is eligible for the study.

Phase 2 (intervention phase). Each subject will be randomly allocated to HD+HP(HA130 once per week) group ,HD+HP(HA330 once per week) group and HD group. The follow-up duration was 3 months.

DETAILED DESCRIPTION:
All patients recruited from these centers who met the inclusion criteria were randomly allocated to HD+HP(HA130 once per week) group ,HD+HP(HA330 once per week) group and HD group. The follow-up duration was 3 months.

Hemoperfusion is performed by HA130 or HA330 resin adsorbents. Blood flow is 200ml/min，dialysate flow is 500ml/min， hemodialysis and hemoperfusion last for 2.5h，continue HD after removing the adsorbent to complete 4 hours'treatment.Heparin for anticoagulation ：first pulse 0.5-1mg/kg ，appending 8-10mg/h. Primary endpoint is the improvement of the clinic symptoms, meanwhile secondary endpoint is serum β2MG、iPTH、CRP、ADMA、BMP2 decrease compared with the baseline, life quality, nutrition condition, and cardiovascular (CVD) incidence.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Stable haemodialysis treatment for more than 3 months, undergoing 2 to 3 times haemodialysis a week for 4 to 5 hours per session
* middle or large molecules retention defined as immunoreactive parathyroid hormone (iPTH) > 400 pg/mL, β2MG>5000 pg/ml、CRP>10mg/l.
* Refractory pruritus, carpal tunnel syndrome, restless leg syndrome, hyperparathyroidism or other refratory complications.

Exclusion Criteria:

* Incapable or reluctant to sign the informed consent or comply the schedule.
* platelet (PLT) count<60×109/L or disturbance in coagulation, tendency of severe bleeding or acute bleeding.
* Severe hypotension and heart or lung insufficiency
* Known hypersensitive or contradiction or intolerance to dialyzer or adsorbents
* Attend to other clinic trial now or in recent 30 days

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
the longitudinal changes of itching | every week, up to 12 weeks.

SECONDARY OUTCOMES:
the longitudinal changes of serum middle molecules of β2MG concentrations | every week,up to 12 weeks.
  The serum concentration of β2MG will be measured using ELISA method
the longitudinal changes of serum middle molecules of iPTH concentrations | every week,up to 12 weeks.
  The serum concentration of iPTH will be measured using ELISA method
the longitudinal changes of serum middle molecules of CRP concentrations | every week,up to 12 weeks.
  The serum concentration of CRP will be measured using ELISA method
the longitudinal changes of serum middle molecules of ADMA concentrations | every week,up to 12 weeks.
  The serum concentration of ADMA will be measured using ELISA method
the longitudinal changes of serum middle molecules of BMP2concentrations | every week,up to 12 weeks.
  The serum concentration of BMP2 will be measured using ELISA method
the longitudinal changes of the nutritional status | every week,up to 12 weeks.
  The nutritional status was evaluated using the serum level of albumin, the subjective global assessment score and BMI. The serum level of albumin will measured using the blood analysis biochemical analyzer, the subjective global assessment score will measured using the SGA scale and the BMI will measured through the physical examination and calculated by weight (kg)/height2 (m2).

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University; Zhihua Zheng, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University; Xunhua Zheng, master, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264